CLINICAL TRIAL: NCT02316340
Title: Modulation of Autophagy: A Clinical Study of Vorinostat Plus Hydroxychloroquine Versus Regorafenib in Refractory Metastatic Colorectal Cancer (mCRC) Patients (CTMS# 14-2015)
Brief Title: Vorinostat Plus Hydroxychloroquine Versus Regorafenib in Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Sukeshi Patel, Principal Investigator, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTMS 14-2015
Record Dates: First submitted 2014-12-09; First posted 2014-12-12 (Estimated); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Vorinostat; Hydroxychloroquine; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Arm - VOR with HCQ (Experimental): Patients will be given vorinostat 400 mg daily and hydroxychloroquine 600 mg daily in 4 week cycles.
  Interventions: Drug: Vorinostat; Drug: Hydroxychloroquine
- Control Arm - Regorafenib (Active Comparator): Patients will be given oral RGF 160 mg daily for 3 weeks in 4 week cycles.
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Vorinostat — 400mg by mouth daily
  Other Names: Zolinza; SAHA; VOR
  Arms: Study Arm - VOR with HCQ
Drug: Hydroxychloroquine — 600mg by mouth daily
  Other Names: HCQ; plaquenil
  Arms: Study Arm - VOR with HCQ
Drug: Regorafenib — 160 mg by mouth daily
  Other Names: Stivarga; RGF
  Arms: Control Arm - Regorafenib

SUMMARY:
This will be a randomized phase II clinical trial of patients with histologic documentation of metastatic colorectal cancer, who have received local and currently approved standard therapies, excluding RGF.

DETAILED DESCRIPTION:
The investigators will give VOR 400 mg PO daily and HCQ 600 mg PO daily in 4-week cycles. Patients will require imaging up to 6 weeks prior to enrollment and will be assessed for measureable evidence of mCRC. This will be a randomized, controlled phase II clinical trial of patients with histological documentation of metastatic colorectal cancer, who have received locally and currently approved standard therapies, excluding RGF. Patients will be randomized 1:1 to RGF or VOR/HCQ (see schema below). Also, crossover is optional after first progression on the initial therapy, and based on physician discretion and in the best interest of the patient. If crossover is not done, then the patient will be off study and can go on to receive other treatments.

ELIGIBILITY:
Inclusion Criteria:

* Histological documentation of metastatic colorectal cancer (mCRC)
* ECOG performance status of 0-2
* Radiographical documentation of metastatic disease with imaging up to 6 weeks prior to enrollment
* Patients with mCRC must have been previously treated with irinotecan and/or oxaliplatin and/or VEGF/EGFR therapy or intolerant to these agents
* Documentation of K-Ras mutational status
* Adequate hematologic, renal and liver function (i.e. absolute neutrophil count > 1000/mm3, platelets > 75,000/mm3); creatinine < 2 times the upper limits of normal (ULN) total bilirubin < 1.5 mg/dl, ALT and AST< 3 times above the ULN, ALT and AST can be < 5 times ULN if patients have hepatic involvement.
* Able to provide written informed consent
* Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception. Women of childbearing potential must have a negative pregnancy test within 72 hours prior to receiving the investigational product
* Tumor blocks available from previous surgery/biopsy, or if not available, patients willing to have biopsy

Exclusion Criteria:

* Patients receiving prior therapy with RGF, VOR, and/or HCQ
* Patients with uncontrolled brain metastases. Patients with brain metastases must be asymptomatic and off corticosteroids for at least one week
* Due to risk of disease exacerbation, patients with porphyria are not eligible
* Due to risk of disease exacerbation, patients with psoriasis are ineligible unless the disease is well controlled, and they are under the care of a specialist for the disorder who agrees to monitor the patient for exacerbations
* Patients with previously documented macular degeneration or diabetic retinopathy
* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study. For targeted therapies, patients will need to clear for 5 half-lives
* Patients may not be receiving any other investigational agents
* Patients should not have taken valproic acid or another histone deacetylase inhibitor for at least 2 weeks prior to enrollment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to VOR or HCQ
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Major surgery or significant traumatic injury occurring within 21 days prior to treatment
* QTc > 500 ms at baseline (average of 3 determinations at 10 minutes interval)
* Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease. Patients with NG-tube, J-tube, or G-tube will not be allowed to participate
* Pregnant women are excluded from this study because vorinostat has the potential for teratogenic or abortifacient effects. For this reason, women of childbearing potential and men must also agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation
* Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with vorinostat, breastfeeding should be discontinued
* Informed Consent - No study specific procedures will be performed without a written and signed informed consent document. Patients who do not demonstrate the ability to understand or the willingness to sign the written informed consent document will be excluded from study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sukeshi Patel Arora, MD, Principal Investigator — University of Texas Health Science Center at the Cancer Therapy and Research Center
Locations (1):
- Cancer Therapy and Research Center University of Texas Health Science Center San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Derived] Arora SP, Tenner L, Sarantopoulos J, Morris J, Liu Q, Mendez JA, Curiel T, Michalek J, Mahalingam D. Modulation of autophagy: a Phase II study of vorinostat plus hydroxychloroquine versus regorafenib in chemotherapy-refractory metastatic colorectal cancer (mCRC). Br J Cancer. 2022 Oct;127(6):1153-1161. doi: 10.1038/s41416-022-01892-6. Epub 2022 Jun 23. PMID 35739299

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were randomized to treatment for the first progression, but crossover was optional after the first progression on the initial therapy and based on physician discretion and in the best interest of the patient. For efficacy analysis: completed at least cycle 1.
Pre-assignment Details: Randomized, controlled trial of VOR 400 mg and HCQ 600 mg PO daily vs RGF 160 mg PO daily (3 weeks on, 1 week off), Q4weeks, in advanced CRC patients. Crossover was optional after first progression.
Period: First Progression
Arm/Group | Study Arm - VOR With HCQ | Control Arm - Regorafenib
Started | 20 | 22
Completed | 17 | 21
Not Completed | 3 | 1
Not completed — Clinical progression | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: Optional Cross-over (MD Discretion)
Arm/Group | Study Arm - VOR With HCQ | Control Arm - Regorafenib
Started | 5 (Efficacy analysis was completed after Cycle 1, crossover was optional, and if not done, then the patient is off the study and can go on to receive other treatments. 13 subjects crossed over to the VOR/HCQ arm) | 13 (Efficacy analysis was completed after Cycle 1. Cross-over was optional, and if not completed then the patient was off-study and could go on to receive other treatments. 5 subjects crossed over to the RGF arm.)
Completed | 2 | 4
Not Completed | 3 | 9

BASELINE CHARACTERISTICS:
Groups:
- Vorinostat/Hydroxychloroquine (VOR/HCQ): Subjects randomized to the VOR/HCQ arm
- Regorafenib (RGF): subjects randomized to the RGF arm
- Total: Total of all reporting groups
Arm/Group | Vorinostat/Hydroxychloroquine (VOR/HCQ) | Regorafenib (RGF) | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Continuous [Median (Full Range); unit: Years] | 58.5 [51.7 to 64] | 57.1 [49.2 to 63] | 58.4 [34.1 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 10 | 17 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 13 | 25
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 22 | 42
Primary location of disease [Count of Participants; unit: Participants]
  Colon | 15 | 15 | 30
  Rectum | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Based on Progression Free Survival of Vorinostat and Hydroxychloroquine Compared to Regorafenib
Description: CT Scan performed every 8 weeks to monitor progression for one year.
Time Frame: Baseline to 12 months
Population: Primary endpoint: median progression-free survival (mPFS) at interim analysis after at least cycle one was completed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Study Arm - VOR With HCQ | Control Arm - Regorafenib
Number analyzed (Participants) | 17 | 21
months | 1.9 [1.87 to 4.35] | 4.35 [1.6 to NA] — not reached

2. Secondary Outcome: Median Overall Survival (mOS)
Description: Overall survival was measured in months from baseline
Time Frame: Baseline up to 22 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Study Arm - VOR With HCQ | Control Arm - Regorafenib
Number analyzed (Participants) | 20 | 22
Months | 6.77 [4.0 to NA] — The CI upper range was undefined due to insufficient number of participants with events | 7.23 [4.8 to 10.8]

ADVERSE EVENTS:
Time Frame: Data collected from baseline up to 22 months.
Groups:
- Study Arm - VOR With HCQ: All study participants that enrolled and were randomized to the study intervention
- Control Arm - Regorafenib: All study participants that enrolled and were randomized to the study control
Arm/Group | Study Arm - VOR With HCQ | Control Arm - Regorafenib
All-Cause Mortality (participants affected / at risk) | 20/20 | 22/22
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/22
Other Adverse Events (participants affected / at risk) | 7/20 | 8/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm - VOR With HCQ (N=20) | Control Arm - Regorafenib (N=22)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bilirubin increased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Elevated transaminases (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hand Foot Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT02316340/Prot_SAP_000.pdf